CLINICAL TRIAL: NCT00228007
Title: Maintaining HIV Risk Reduction Among Needle Exchangers
Brief Title: Antidepressant Medication for Reducing HIV Risk Behavior in Depressed Intravenous Drug Users
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Michael Stein, M.D./Principal Investigator, RI Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH062719 (NIH); R01MH062719 (NIH); DAHBR AZ-Q
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Depression; Substance-Related Disorders; HIV Infections
Keywords: Injection Drug Use; HIV Risk Behavior; HIV Seronegativity
MeSH Terms: conditions — Depression; Substance-Related Disorders; HIV Infections | interventions — Antidepressive Agents

INTERVENTIONS:
Drug: Antidepressant Medication

SUMMARY:
This study will evaluate the effectiveness of antidepressant medication treatment in reducing HIV risk behaviors in intravenous drug users with depression.

DETAILED DESCRIPTION:
Depression and injection drug use often come hand-in-hand. This is especially true in populations with limited access to mental health care and with a high risk of illness and HIV transmission. Depressed injection drug users in these populations usually continue their drug use for extended periods of time, thereby further promoting the spread of HIV. This cycle has created a significant public health problem. It is necessary to explore new approaches to facilitate and maintain long-term behavior changes within this population. This study will evaluate the effectiveness of treatment with antidepressant medications in reducing HIV risk behaviors in depressed intravenous drug users.

Participants in this open label study will be randomly assigned to receive either antidepressant treatment or no treatment. Participants in the treatment group will meet with a psychiatrist monthly for 12 months. Based on psychiatric evaluations and participants' medical histories, doctors will prescribe an appropriate antidepressant medication or a combination of medications. Participants in the treatment group may also receive referrals for other services if necessary. Participants assigned to receive no treatment will be contacted at Months 3 and 9 to verify their contact information; they will also receive any necessary referrals. All participants will partake in interviews at baseline and Months 6 and 12 to assess changes in HIV risk behavior and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depression, dysthymia, substance-induced major depression, or major depression plus dysthymia
* Score of greater than 14 on the Hamilton Rating Scale for Depression
* Current opiate or cocaine use
* History of injection equipment sharing
* English-speaking

Exclusion Criteria:

* History of injection equipment sharing within 6 months of study entry
* Currently at risk for suicide
* Currently experiencing symptoms of psychosis
* Currently taking any other psychotropic medication
* Diagnosed with bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, or paranoid disorder
* Informed that treatment with antidepressant medications is medically inadvisable
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265
Dates: Start 2000-09; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Maintenance of HIV risk-free drug behavior (measured at Month 12)

SECONDARY OUTCOMES:
Reduction in depressive symptoms (measured at Month 12)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Rhode Island Hospital; Penelope Dennehy, MD, Study Director — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Hayaki J, Stein MD, Lassor JA, Herman DS, Anderson BJ. Adversity among drug users: relationship to impulsivity. Drug Alcohol Depend. 2005 Apr 4;78(1):65-71. doi: 10.1016/j.drugalcdep.2004.09.002. PMID 15769559